CLINICAL TRIAL: NCT02926261
Title: Evaluation of Three Methods for Nutritional Assessment in Patients With Cirrhosis
Brief Title: Methods for Nutritional Assessment in Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, MD, MSc, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: BIVA0978
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-01

CONDITIONS: Liver Cirrhosis; Cachexia; Malnutrition
MeSH Terms: conditions — Liver Cirrhosis; Cachexia; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma samples collected at time of evaluation and stored at -80°.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Bioelectrical impedance vector analysis — Evaluation of nutritional status with Bioelectrical impedance vector analysis, hand-grip strength and computed-tomography scan

SUMMARY:
Nutritional status in patients with cirrhosis has been shown to have a direct influence on the prognosis of these patients, it is related to higher mortality and it has been linked to the developement and perpetuation of certain complications such as hepatic encephalopathy, ascites and spontaneous bacterial peritonitis.

Despite the importance of nutritional status in this patients, most of the methods for its assessment are still not completely reliable or not easily accessible; therefore, evaluating nutritional status in the daily clinical practice is still a complex task.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis
* No restriction of etiology
* 18-75 years
* Child-Pugh stage A/B/C
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Extremity amputation
* Malignancy different from hepatocellular carcinoma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patients with cirrhosis
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | Evaluation at time of recruitment
  Characterization of nutritional status by three methods of nutritional assessment
  * Bioelectrical impedance vector analysis
  * CT scan
  * Handgrip strength

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre, MD, MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No